CLINICAL TRIAL: NCT07039877
Title: Efficacy of Low-dose Venetoclax With Itraconazole + TACL in Patients With Relapsed/Refractory Acute Lymphoblastic Leukemia
Brief Title: Efficacy of Low-dose Venetoclax With Itraconazole + TACL for R/R ALL Patients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hospital Universitario Dr. Jose E. Gonzalez (Other)
Responsible Party: Principal Investigator, David Gomez Almaguer, Head of Hematology, Hospital Universitario Dr. Jose E. Gonzalez
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HE25-00004
Record Dates: First submitted 2025-06-18; First posted 2025-06-26 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Acute Lymphobkastic Leukemia; Acute Lymphoblastic Leukaemia Recurrent; Philadelphia Chromosome Negative ALL
Keywords: ALL; relapsed ALL; Venetoclax; TACL; refractoy ALL
MeSH Terms: interventions — venetoclax; Itraconazole

STUDY DESIGN:
Intervention Model Description: One arm, open-label, phase 2 study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TACL plus low dose Venetoclax and Itraconazole (Experimental): Salvage chemotherapy will be assigned as follows:
  * Venetoclax 100 mg orally every day for 7 days
  * Itraconazole 100 mg orally every 12 hours for 7 days
  * Vincristine 1.4 mg/m2 intravenously on days 1, 8, 15, and 22
  * Mitoxantrone 6 mg/m2 intravenously on day 1
  * L-Asparaginase 6,000 IU/m2 intramuscularly on days 5, 7, 9, 11, 13, 16, 18, 20, and 23
  * Dexamethasone 16 mg orally from days 1 to 15
  * Bortezomib 2 mg subcutaneously on days 1, 4, 8, and 11
  * Rituximab 375 mg/m2 intravenously on day 8 for patients with CD20+, more than 20% expression
  * Intrathecal Chemotherapy or CNS (-): Days 8 and 15 or CNS (+): Days 1, 8, 15, and 22
  Interventions: Drug: Venetoclax low dose with itraconazole

INTERVENTIONS:
Drug: Venetoclax low dose with itraconazole — The investigators will add venetoclax in low dose (100 mg) with itraconazole to the pediatric inspired regimen TACL to enchance the complete response rate

SUMMARY:
Relapsed/refractory acute lymphoblastic leukemia remains a challenge in the context of limited access to immunotherapy in developing countries. With such poor 5-year overall survival rates of 10%, the investigators need strategies that surpass the complete response rate achieved in this setting, which does not exceed 60% effectiveness with different regimens, and to eventually transfer patients to hematopoietic stem cell transplantation.

In this context, the investigators are studyng if the use of venetoclax, a BCL2 inhibitor, with the use of a cytochrome p450 inhibitor such as itraconazole, alongside the TACL chemotherapy regimen, which is based on the combination of asparaginase, dexamethasone, bortezomib, vincristine, and mitoxantrone.

DETAILED DESCRIPTION:
Response rates for salvage regimens vary depending on the patient's performance status (suitable or unsuitable for high-intensity chemotherapy), whether the patient is refractory (40%), in early or late first relapse (up to 60%), and in second or later relapse, where complete response rates decrease dramatically (as low as 10% with high-intensity regimens). Post-refractory OS has been reported at 5 months, with an EFS of 4.7 months. For patients in first relapse, the reported studies range from 5.8 months for those receiving salvage chemotherapy alone, increasing to 10 months if they undergo hematopoietic progenitor cell transplantation. For second relapses or relapses after transplantation, OS does not exceed 5 months. For patients who do not receive any treatment, the prognosis is grim, with high mortality within the following months following refractoriness or relapse without any support. 30,31,32

Therefore, it is proposed to increase the complete response rate with a pediatric-inspired chemotherapy regimen in conjunction with a BCL-2 inhibitor, so that patients can be transitioned to allogeneic bone marrow transplantation (the only curative therapy in this context), either after the treatment received or with short-term immunotherapy bridging to transplantation.

The risks associated with conventional salvage chemotherapy for patients with good performance status will not differ significantly from those typically observed in daily clinical practice (see below for the expected description of adverse events), since the basis of therapy remains the TACL regimen. A higher degree of cytopenias, especially neutropenia and thrombocytopenia, can be expected with the addition of a BCL-2 inhibitor.

Salvage chemotherapy will be assigned as follows:

* Venetoclax 100 mg orally every day for 7 days
* Itraconazole 100 mg orally every 12 hours for 7 days
* Vincristine 1.4 mg/m2 intravenously on days 1, 8, 15, and 22
* Mitoxantrone 6 mg/m2 intravenously on day 1
* L-Asparaginase 6,000 IU/m2 intramuscularly on days 5, 7, 9, 11, 13, 16, 18, 20, and 23
* Dexamethasone 20 mg orally from days 1 to 15
* Bortezomib 2 mg subcutaneously on days 1, 4, 8, and 11
* Rituximab 375 mg/m2 intravenously on day 8 for patients with CD20+, more than 20% expression in flow cytometry
* Intrathecal Chemotherapy or CNS (-): Days 8 and 15 or CNS (+): Days 1, 8, 15, and 22

The proposed chemotherapy regimen will be administered orally, intravenously, intramuscularly, and subcutaneously in an outpatient setting on the previously specified days, with appointments scheduled on days 1, 8, 15, and 22 for drug administration on the fifth floor of the University Cancer Center in the Hematology Service area. General patient assessment will be conducted in the ground floor offices of the University Cancer Center's Hematology Service. Any adverse events will be reported by system and grade according to CTCAE.

After completing the salvage chemotherapy regimen, bone marrow aspiration and measurable residual disease will be assessed on day 29 of the cycle, and not beyond day 35.

ELIGIBILITY:
Inclusion Criteria:

* B-cell or T-cell acute lymphoblastic leukemia.
* Philadelphia chromosome negative
* Relapsed disease after any line of treatment, defined as detection of disease activity at any time after remission
* Refractory disease after first-line treatment, defined as: more than 5% blasts after completion of induction/consolidation by flow cytometry
* Not having included venetoclax in any prior regimen.
* No prior organ damage, defined as the absence of any serious, life-threatening disease prior to the start of treatment.
* Performance status defined by the ECOG scale between 0 and 2.

Exclusion Criteria:

* Isolated CNS relapse.
* Performance status defined by ECOG scale between 3 and 4.
* CTCAE-classified sensory or motor neuropathy of grade 3 or higher.
* History of hypersensitivity or intolerance to the drugs included in the regimen.
* Prior organ damage, defined as the presence of any serious, life-threatening illness prior to the start of treatment.

Ages: 16 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-01-02 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Overall response rata after low dose venetoclax with itraconazole plus TACL | 16 months
  To evaluate the overall response after reinduction to remission with low dose venetoclax plus TACL in patients with relapsed/refractory acute lymphoblastic leukemia

SECONDARY OUTCOMES:
Percentage of measurable residual disease in complete response | 16 months
  Describe the percentage of residual measurable disease in patients with complete response or complete response with incomplete hematologic recovery
Adverse events evaluatio | 16 months
  Identify the most frequent adverse events following the administration of venetoclax + TACL according to the CTCAE version 5 criteria
Patients recieving HSCT after chemotherapy | 24 months
  Determinate the percentage of patients who receive hematopoietic stem cell transplant after treatment with low dose venetoclax with itraconazole plus TACL
Event-free survival | 24 months
  Evaluate event-free survival following low dose venetoclax with itraconazole plus TACL regimen
Overall survival | 24 months
  Evaluate overall survival following low dose venetoclax with itraconazole plus TACL regimen

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Dr. Jose E. Gonzalez, Monterrey, Nuevo León, Mexico

REFERENCES:
- [Background] Colunga-Pedraza JE, Gonzalez-Llano O, Gonzalez-Martinez CE, Gomez-Almaguer D, Yanez-Reyes JM, Jimenez-Antolinez V, Colunga-Pedraza PR. Outpatient low toxic regimen with bortezomib in relapsed/refractory acute lymphoblastic leukemia in pediatrics and AYA patients: Single-center Mexican experience. Pediatr Blood Cancer. 2020 May;67(5):e28241. doi: 10.1002/pbc.28241. Epub 2020 Mar 11. PMID 32159276